CLINICAL TRIAL: NCT00108576
Title: Divalproex Sodium in the Treatment of PTSD: A Placebo-Controlled Study
Brief Title: Divalproex Sodium in the Treatment of PTSD (Post-Traumatic Stress Disorder)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBS-026-01
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: PTSD
Keywords: anticonvulsant; anxiety; divalproex; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): Look-a-like placebo
  Interventions: Other: placebo
- Arm 2 (Experimental): Divalproex
  Interventions: Drug: Divalproex

INTERVENTIONS:
Drug: Divalproex — anticonvulsant; mood stabilizer
  Arms: Arm 2
Other: placebo — Look-a-like placebo
  Arms: Arm 1

SUMMARY:
The purposes of this study are:

* To study the efficacy of divalproex in the treatment of PTSD;
* To study the plasma GABA (gamma aminobutyric acid) levels before and after treatment with divalproex in PTSD.

DETAILED DESCRIPTION:
Objective: To study the efficacy of divalproex in the treatment of PTSD. Research Design: This is an 8-week randomized, double-blind, placebo-controlled treatment trial of divalproex.

Methodology: After signing an informed consent and meeting all inclusion/exclusion criteria, the patient is randomized to either divalproex or placebo for an 8-week duration. During the study a pharmacist maintains the randomization log and administers the placebo or divalproex (500 mg/capsule) in look-a-like tablets. Patients' symptoms, side effects and compliance are assessed bi-weekly. Based on symptomology and occurrence of side effects, the investigator increases the medication in 500 mg (one tablet) increments every four days, as tolerated, until a maximum therapeutic benefit is achieved, not to exceed 3000 mg/day (6 capsules). The dosing is twice daily, with the higher dose at bedtime. Compliance is assessed by bi-weekly pill count and blinded valproic acid levels at week 4 and week 8. Patients are given supportive clinical management during the clinic visits. An investigator is available by telephone 24 hrs a day in case of emergency. Patients may be seen more often if needed. Efficacy will be measured by the following assessment scales: MADRS (Montgomery-Asberg Depression Rating Scale), Ham-A (Hamilton Anxiety Scale), CGI-s (Clinical Global Impressions-Severity of Illness Scale), CGI-I (Clinical Global Impressions-Improvement Scale), GAF (Global Assessment of Functioning), CAPS (Clinician-Administered PTSD Scale), TOP-8 (Treatment Outcome PTSD Rating Scale), and DTS (Davidson Trauma Scale). Results of this study will be used to evaluate the efficacy of divalproex in the treatment of PTSD.

Significance: Divalproex has shown promise in treating PTSD in open label trials. This study is the next step in proving divalproex's efficacy in the treatment of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD, confirmed by MINI (Mini-International Neuropsychiatric Interview) and CAPS
* Age 19 or older
* No substance abuse/dependence for the previous 6 weeks (except for nicotine and caffeine)
* Free of psychotropic medication for 2 weeks (except 6 weeks for fluoxetine)
* Clinically normal physical and laboratory examination (lab profile listed below). LFTs (liver function tests) up to 2.5 times the normal limit will be allowed.
* Women of childbearing potential must be using medically approved methods of birth control (such as a condom, birth control pill, Depo-Provera, or diaphragm with spermicides)
* Signed informed consent
* Male or female of any race or ethnic origin

Exclusion Criteria:

* Lifetime history of bipolar I, psychotic, or cognitive disorders
* Actively suicidal, homicidal, or psychotic
* History of sensitivity to divalproex
* Unstable general medical conditions
* Score 6 on Question #10 of MADRS
* Women who are pregnant, planning to become pregnant or to breastfeed during the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2003-10; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lynne Davis, MD AB, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

REFERENCES:
- [Derived] Davis LL, Davidson JR, Ward LC, Bartolucci A, Bowden CL, Petty F. Divalproex in the treatment of posttraumatic stress disorder: a randomized, double-blind, placebo-controlled trial in a veteran population. J Clin Psychopharmacol. 2008 Feb;28(1):84-8. doi: 10.1097/JCP.0b013e318160f83b. PMID 18204347